CLINICAL TRIAL: NCT01569711
Title: Preliminary Study Evaluating Deep Brain Stimulation of Nucleus Accumbens in Patients Suffering From Chronic and Resistant Major Depressive Disorder
Brief Title: Deep Brain Stimulation of Nucleus Accumbens for Chronic and Resistant Major Depressive Disorder
Acronym: PRESTHYM
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-A00234-51
Record Dates: First submitted 2012-02-24; First posted 2012-04-03 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Major Depressive Disorder, Recurrent, Unspecified
Keywords: chronic and resistant major depressive disorder; deep brain stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deep brain stimulation
  Interventions: Procedure: Deep brain stimulation of nucleus accumbens

INTERVENTIONS:
Procedure: Deep brain stimulation of nucleus accumbens — * Day0 : surgical placement of electrodes
  * M1 : stimulation of nucleus accumbens
  * M5 : stimulation of nucleus accumbens or associative territory of caudate nucleus (if no response observed with nucleus accumbens stimulation)
  Other Names: Non applicable.

SUMMARY:
Depression is a common, recurrent and disabling disorder. Among patients with a chronic course of the disease, 20 to 30% are resistant to antidepressant medications. Among those patients, 50% would not benefit from electroconvulsive therapy (ECT). For such patients, deep brain stimulation (DBS) of nucleus accumbens is considered.

DETAILED DESCRIPTION:
Depression is a common (12-Month Prevalence in the general population: 6%), recurrent and disabling disorder.

Among patients with a chronic course of the disease, 20 to 30% are resistant to antidepressant medications. Among those patients not responding favorably to antidepressant medications, 50% would not benefit from ECT. For such patients, surgical interventions have been proposed in the past.

Many results support the hypothesis of a dysfunction of the functional loops between cortical and subcortical structures underlying the expression of depressive disorders.

Thus, therapeutic intervention focusing on these loops, in patients with chronic depression resistant to treatment, should be an issue and could improve prognosis of these patients.

As part of a maximal resistance to antidepressant drug, after failure of a series of bilateral ECT, a surgical functional intervention using DBS of nucleus accumbens is considered.

This open-label trial proposes to assess feasibility, safety and efficacy of DBS of nucleus accumbens in patients with chronic depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 30 and 60 years old
* Meeting DSM-IV-TR for a major depressive disorder (MDD), recurrent (296.3x) diagnosed using the MINI scale
* Duration of the episode > 2 years
* History of recurrent MDD (at least one prior episode index), authenticated by a report of ambulatory care or hospitalization
* Meeting Thase and Rush stage V for resistance (Thase and Rush 1997) (Annex 1 : mettre l'annexe)
* Presenting simultaneously an HDRS total score (17 items)> 21, a GAF <50, and a score of 4 on CGI despite the use of all the following strategies :

  * monotherapy: 2 SSRIs, 1 ISRNA, 1 tricyclic (with measurement of plasma) at the maximum prescribed for a period of 8 weeks
  * association at least one previous antidepressant, and for at least six weeks of one of the following treatment: lithium, thyroid hormone, buspirone, pindolol. An intolerance to one of these drug treatments related to its known side effects will be considered equivalent to the lack of effect of this treatment
  * irreversible MAOI: iproniazid (Marsilid *)
  * combination of 2 antipsychotics, with at least a second generation antipsychotic (olanzapine, risperidone, amisulpride, aripiprazole or clozapine)
  * combination of 2 antidepressants
  * ECT: at least 8 sessions in maximal load with crisis GET> 25 sec bilaterally. If not possible by cognitive impairment: unilateral
  * structured psychotherapy inspired cognitive-behavioral or other type of structured psychotherapy for a period of one year
* Understanding of the study
* Giving their written, free and informed consent
* Affiliated to social security

Exclusion Criteria:

* Serious and unstable medical condition (cardiovascular, respiratory, endocrine, metabolic, liver, renal, hematologic, infectious, neurological or other ...) making impossible the establishment of study treatment
* Cognitive deterioration (Mattis < 130)
* Abnormal brain standard MRI or contraindication for MRI
* Axis 1 disorder other than MDD (except generalized anxiety disorder, social phobia, panic disorder)
* Addiction to alcohol and other psychoactive substances with the exception of nicotine
* suicide risk in the last month (MINI 5.0.0: section suicide risk DIGS: section intent, premeditation, lethality) and score> 2 in item 3 of HDRS
* More than two suicide attempts within two years prior to inclusion
* MDD with psychotic features congruent or incongruent to the mood or an history of MDD with psychotic features
* Diagnostic criteria for personality disorders according to DSM-IV-TR Cluster A or B evaluated using the SCID2 (Maffei et al., 1997)
* Involuntary commitment, guardianship or trusteeship
* Women of childbearing without effective contraception

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a chronic and resistant major depressive disorder.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
response after four months (M5) of DBS months defined as a 50% decrease in HDRS score | At 5 months after the DBS
  The primary outcome is response after four months (M5) of DBS months defined as a 50% decrease in HDRS score.

SECONDARY OUTCOMES:
Remission (defined as a score in the HDRS ≤ 7) after 4 months | At 5 months after the DBS
Duration of remission in the year of postoperative follow-up | at one year of postoperative follow-up
Obtaining an overall score on the scale Anxiety Hamilton (HARS) ≤ 10 during the year of postoperative follow-up | at one year of postoperative follow-up
Getting a score from 1 ("very much improved") or 2 ("strongly improved ") to item 2 of the Clinical Global Impression (CGI) during the year of postoperative follow-up | at one year of postoperative follow-up
Obtaining a score ≥ 60 at the level of Global Assessment of Functioning (GAF) during the year of postoperative follow-up | at one year of postoperative follow-up
Changes in score on the scale of social adjustment in its self-assessment by (SAS-SR) in the year of postoperative follow-up | at one year of postoperative follow-up
Evaluation of tolerance to treatment by clinicians, and by the patient and his family circle, reporting by the patient for adverse events at each follow-up visits after surgery, completion of the initial neuropsychological checkup | at each follow-up visits after surgery
Effect of DBS at M9 after the DBS on caudate nucleus in case of non response at M5 after the DBS. | at 9 months after the DBS
  The same scales (as described before) will be used at M9, to describe the effect of DBS on caudate nucleus.

CONTACTS AND LOCATIONS:
Overall Officials: Millet MD Bruno, Principal Investigator — Rennes University Hospital
Locations (10):
- France (10):
  - Grenoble University Hospital (Nord Hospital), Grenoble, France
  - Bordeaux UH, Bordeaux
  - Gabriel montpied University Hospital, Clermont-Ferrand
  - Lille UH (Roger Salengro Hospital), Lille
  - Lyon UH (Pierre Wertheimer Hospital), Lyon
  - La Salpétrière UH, Paris
  - Sainte Anne UH, Paris
  - Poitiers UH, Poitiers
  - Rennes UH, Rennes
  - Toulouse UH, Toulouse

REFERENCES:
- [Derived] Millet B, Jaafari N, Polosan M, Baup N, Giordana B, Haegelen C, Chabardes S, Fontaine D, Devaux B, Yelnik J, Fossati P, Aouizerate B, Krebs MO, Robert G, Jay T, Cornu P, Verin M, Drapier S, Drapier D, Sauleau P, Peron J, Le Jeune F, Naudet F, Reymann JM. Limbic versus cognitive target for deep brain stimulation in treatment-resistant depression: accumbens more promising than caudate. Eur Neuropsychopharmacol. 2014 Aug;24(8):1229-39. doi: 10.1016/j.euroneuro.2014.05.006. Epub 2014 May 20. PMID 24950819